CLINICAL TRIAL: NCT00678288
Title: A Phase II, Randomized, Open-label, Multicenter, Study Evaluating the Efficacy of Sorafenib Alone and Sorafenib in Combination With Low Dose Interferon Alpha-2a as Second-line Treatment of Sunitinib Failure in Patients With Metastatic Renal Cell Carcinoma
Brief Title: A Study to Assess Sorafenib Alone and in Combination With Low-Dose Interferon Following Unsuccessful Treatment With Sunitinib in Patients With Advanced Renal Cell Cancer.
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 12782; 2007-005083-28 (EudraCT Number); CONCERT (Other: Bayer)
Record Dates: First submitted 2008-05-14; First posted 2008-05-15 (Estimated); Results first posted 2010-10-01 (Estimated); Last update posted 2014-12-11 (Estimated); Status verified 2014-11

CONDITIONS: Carcinoma, Renal Cell
Keywords: Renal Cell Cancer; Interferon
MeSH Terms: conditions — Carcinoma, Renal Cell | interventions — Sorafenib; Interferons

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sorafenib (Nexavar, BAY43-9006) (Experimental): Sorafenib 400 mg (two 200 mg tablets) twice daily (bid) per os (po), continuously.
  Interventions: Drug: Sorafenib (Nexavar, BAY43-9006)
- Sorafenib (Nexavar, BAY43-9006) + Interferon (Experimental): Sorafenib 400 mg (two 200 mg tablets) twice daily (bid) per os (po), continuously plus Interferon (IFN) alpha-2a 3 millions of international unit (MIU) five times a week (FIW) subcutaneous (s.c.), from Monday to Friday (total weekly dose 15 MIU) s.c., to start one week after commencing sorafenib.
  Interventions: Drug: Sorafenib (Nexavar, BAY43-9006) + Interferon

INTERVENTIONS:
Drug: Sorafenib (Nexavar, BAY43-9006) — Sorafenib 400 mg (two 200 mg tablets) BID PO, continuously
  Arms: Sorafenib (Nexavar, BAY43-9006)
Drug: Sorafenib (Nexavar, BAY43-9006) + Interferon — Sorafenib 400 mg (two 200 mg tablets) BID PO, continuously. IFN alpha-2a 3MIU FIW s.c., from Monday to Friday (total weekly dose 15 MIU) s.c., to start one week after commencing sorafenib.
  Arms: Sorafenib (Nexavar, BAY43-9006) + Interferon

SUMMARY:
This study is to assess sorafenib as second treatment for patients that have previously received only sunitinib as first-line treatment for advanced renal cell cancer, and who either responded and then progressed with sunitinib or were intolerant to sunitinib. This study is to assess if combining the usual dose of sorafenib (200mg twice-daily) with low dose interferon (3 million international unit (MIU) five times a week) can treat kidney cancer more effectively than the current approved dose alone and if it is safe. In addition, for patients that respond to treatment with sorafenib alone or in combination with interferon before progressing, patients may receive sorafenib alone at an increased dose of 300mg twice-daily, provided that toxicities are acceptable and at the discretion of the investigator.

ELIGIBILITY:
Inclusion Criteria:

* Disease progression as defined by Response Evaluation Criteria in Solid Tumors (RECIST) criteria following documented stable disease or better after at least 8 weeks of sunitinib as first-line treatment (or two cycles of 4 weeks on and 2 weeks off treatment)
* And/or patients who have discontinued sunitinib treatment at any point due to toxicity
* Study entry at least 2 weeks after treatment with sunitinib but up to a maximum of 8 weeks
* Memorial Sloane Kettering Cancer Centre (MSKCC) prognostic score low or intermediate
* Eastern Cooperative Oncology Group (ECOG) Performance Status of 0 or 1
* Patient must have histologically confirmed metastatic renal cell carcinoma with predominant clear cell histology (clear cell component more than 50%).

Exclusion Criteria:

* Patient should be excluded if they have unresolved chronic toxicity grade
* > 1 and related to prior therapy with sunitinib.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2008-04; Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (32):
- Austria (2):
  - Vienna, Vienna
  - Salzburg
- France (10):
  - Avignon
  - Bayonne
  - Bordeaux
  - Marseille
  - Nantes
  - Paris
  - Reims
  - Strasbourg
  - Toulouse
  - Vandœuvre-lès-Nancy
- Ireland (2):
  - Dublin, Dublin
  - Cork
- Italy (6):
  - Aviano, Pordenone
  - Legnago, Verona
  - Napoli
  - Pavia
  - Perugia
  - Reggio Emilia
- Poland (4):
  - Gdansk
  - Lublin
  - Warsaw
  - Wroclaw
- Spain (5):
  - Barcelona, Barcelona
  - Madrid, Madrid
  - Oviedo, Oviedo
  - Pamplona, Pamplona
  - Valencia, Valencia
- United Kingdom (3):
  - London, London
  - Northwood, Middlesex
  - Newcastle upon Tyne, Tyne and Wear

REFERENCES:
- See also: Click here and search for EudraCT infomation of Bayer Product — http://www.clinicaltrialsregister.eu

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted from 16 Apr 2008 to 26 Jun 2009 at 31 centers in 7 countries: France (11), Italy (6), Spain (5), Poland (4), Ireland (2), United Kingdom (2), and Austria (1). The planned enrollment was 120 subjects in the 2 treatment groups (60 subjects per group). The study was stopped early because of slow accrual.
Pre-assignment Details: A total of 24 subjects were screened; 16 were enrolled and randomized; 10 (63%) to sorafenib alone and 6 (37%) to sorafenib + interferon. All 16 randomized subjects received at least 1 dose of study drug and were included in the safety analysis population.
Period: Overall Study
Arm/Group | Sorafenib (Nexavar, BAY43-9006) | Sorafenib (Nexavar, BAY43-9006) + Interferon
Started | 10 | 6
Completed | 0 | 0
Not Completed | 10 | 6
Not completed — Adverse Event | 0 | 2
Not completed — Withdrawal by Subject | 1 | 1
Not completed — Study terminated by the sponsor | 2 | 0
Not completed — Not compliant with study medication | 0 | 1
Not completed — Switch to commercial drug | 0 | 1
Not completed — Reason not reported | 1 | 0
Not completed — Disease progression/recurrence/relapse | 6 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Sorafenib (Nexavar, BAY43-9006) | Sorafenib (Nexavar, BAY43-9006) + Interferon | Total
Number analyzed (Participants) | 10 | 6 | 16
Age, Continuous [Median (Full Range); unit: years] | 57 [41 to 67] | 60.5 [48 to 73] | 58.5 [41 to 73]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 4 | 7
  Male | 7 | 2 | 9
Memorial Sloane Kettering Cancer Center (MSKCC) score [Number; unit: participants] — The MSKCC score is a prognostic score obtained by adding 1 point for each of 5 risk factors: 1. Absence of prior nephrectomy, 2. Corrected serum calcium > 10 mg/dL, 3. Hemoglobin < lower limit of normal, 4. Lactate dehydrogenase (LDH) > 1.5X upper limit of normal, 5. Eastern Cooperative Oncology Group (ECOG) Performance Status (PS) ≥ 2 (The ECOG PS is a scale that measures how cancer affects a patient. The scale ranges from 0 [fully active] to 5 [dead]). A Low MSKCC score is 0 risk factors, Intermediate is 1-2 risk factors, and Poor is 3-5 risk factors.
  participants
    low MSKCC score | 3 | 1 | 4
    intermediate MSKCC score | 7 | 5 | 12

OUTCOME MEASURES:

1. Primary Outcome: Progression-Free Survival
Description: Progression-free Survival (PFS) was the time from the first dose of combination therapy to disease progression (radiological or clinical, whichever is earlier, according to Response Evaluation Criteria in Solid Tumors [RECIST]) or death (if death occurs before progression is documented). PFS for subjects without tumor progression or death at the time of analysis were censored at the date of last tumor evaluation.
Time Frame: From start of treatment of the first subject until 14 months later, assessed every 8 weeks
Population: Efficacy analysis was not performed due to low accrual. For details, please see Limitation and Caveats.
Arm/Group | Sorafenib (Nexavar, BAY43-9006) | Sorafenib (Nexavar, BAY43-9006) + Interferon
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Response Rate
Description: Response Rate was the best tumor response (confirmed Complete Response [CR], Partial Response [PR] or Stable Disease [SD]) observed according to the Response Evaluation Criteria in Solid Tumors (RECIST) criteria.
Time Frame: From start of treatment of the first subject until 14 months later, assessed every 8 Weeks
Population: Efficacy analysis was not performed due to low accrual. For details, please see Limitation and Caveats.
Arm/Group | Sorafenib (Nexavar, BAY43-9006) | Sorafenib (Nexavar, BAY43-9006) + Interferon
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Time to Progression
Description: Time to progression was the time from treatment start date to disease progression. Subjects without progression at the time of analysis were censored at their last date of tumor evaluation.
Time Frame: From start of treatment of the first subject until 14 months later, assessed every 8 Weeks
Population: Efficacy analysis was not performed due to low accrual. For details, please see Limitation and Caveats.
Arm/Group | Sorafenib (Nexavar, BAY43-9006) | Sorafenib (Nexavar, BAY43-9006) + Interferon
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Duration of Response
Description: Duration of Response was the time from date of first response (Complete Response [CR] or Partial Response [PR]) to the date when Progressive Disease (PD) is first documented or to the date of death, whichever occurs first. Subjects still having CR or PR at the time of analysis were censored at their last date of last contact.
Time Frame: From start of treatment of the first subject until 14 months later, assessed every 8 Weeks
Population: Efficacy analysis was not performed due to low accrual. For details, please see Limitation and Caveats.
Arm/Group | Sorafenib (Nexavar, BAY43-9006) | Sorafenib (Nexavar, BAY43-9006) + Interferon
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Overall Survival
Description: Overall Survival was the time from treatment start date to death due to any cause. Subjects still alive at the time of analysis were censored at their last date of last contact.
Time Frame: From start of treatment of the first subject until 14 months later, assessed every 8 Weeks
Population: Efficacy analysis was not performed due to low accrual. For details, please see Limitation and Caveats.
Arm/Group | Sorafenib (Nexavar, BAY43-9006) | Sorafenib (Nexavar, BAY43-9006) + Interferon
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Description: Acronyms in Adverse Event section: not otherwise specified (NOS), Alanine transaminase (ALT), Aspartate transaminase (AST)
Arm/Group | Sorafenib (Nexavar, BAY43-9006) | Sorafenib (Nexavar, BAY43-9006) + Interferon
Serious Adverse Events (participants affected / at risk) | 5/10 | 3/6
Other Adverse Events (participants affected / at risk) | 9/10 | 5/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Sorafenib (Nexavar, BAY43-9006) (N=10) | Sorafenib (Nexavar, BAY43-9006) + Interferon (N=6)
Fatigue (General disorders) | 1 | 2
Infection (documented clinically), bronchus (Infections and infestations) | 1 | 0
Fracture (Musculoskeletal and connective tissue disorders) | 1 | 1
Pain, bone (General disorders) | 1 | 0
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pain, back (General disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Sorafenib (Nexavar, BAY43-9006) (N=10) | Sorafenib (Nexavar, BAY43-9006) + Interferon (N=6)
Rhinitis (Immune system disorders) | 1 | 0
Tinnitus (Ear and labyrinth disorders) | 1 | 0
Neutrophils (Blood and lymphatic system disorders) | 1 | 0
Hemoglobin (Blood and lymphatic system disorders) | 1 | 1
Platelets (Blood and lymphatic system disorders) | 1 | 2
Leukocytes (Blood and lymphatic system disorders) | 1 | 0
Hypertension (Cardiac disorders) | 2 | 0
Fatigue (General disorders) | 7 | 3
Weight loss (General disorders) | 1 | 0
Anorexia (Gastrointestinal disorders) | 2 | 2
Diarrhea (Gastrointestinal disorders) | 5 | 3
Mucositis (functional/symptomatic), esophagus (Gastrointestinal disorders) | 1 | 0
Mucositis (functional/symptomatic), oral cavity (Gastrointestinal disorders) | 2 | 1
Mucositis (functional/symptomatic), pharynx (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 1 | 3
Taste alteration (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 2 | 2
Infection (documented clinically), bronchus (Infections and infestations) | 1 | 0
Infection (documented clinically), dental-tooth (Infections and infestations) | 1 | 0
Dermal change (Skin and subcutaneous tissue disorders) | 1 | 0
Extremity-upper (function) (Musculoskeletal and connective tissue disorders) | 1 | 0
Metabolic/lab - other (Metabolism and nutrition disorders) | 1 | 1
Mood alteration, depression (Nervous system disorders) | 1 | 0
Neuropathy: sensory (Nervous system disorders) | 1 | 1
Pain, back (General disorders) | 1 | 1
Pain, chest/thorax NOS (General disorders) | 2 | 0
Pain, chest wall (General disorders) | 1 | 0
Pain, abdomen NOS (General disorders) | 4 | 0
Pain, head/headache (General disorders) | 1 | 1
Pain, joint (General disorders) | 1 | 0
Pain, bone (General disorders) | 1 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 2 | 2
Voice changes (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 2 | 0
Hand-foot skin reaction (Skin and subcutaneous tissue disorders) | 5 | 0
Dermatology - other (Skin and subcutaneous tissue disorders) | 2 | 0
Photosensitivity (Skin and subcutaneous tissue disorders) | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 1
Rash/desquamation (Skin and subcutaneous tissue disorders) | 5 | 3
Flushing (Skin and subcutaneous tissue disorders) | 2 | 0
Libido (Reproductive system and breast disorders) | 1 | 0
Thrombosis/thrombus/embolism (Vascular disorders) | 1 | 0
Auditory/ear - ohter (Ear and labyrinth disorders) | 0 | 1
Hypothyroidism (Endocrine disorders) | 0 | 1
Fever (General disorders) | 0 | 2
Insomnia (General disorders) | 0 | 1
Constitutional symptoms - other (General disorders) | 0 | 1
Constipation (Gastrointestinal disorders) | 0 | 1
Dehydration (Gastrointestinal disorders) | 0 | 1
Hematoma (Vascular disorders) | 0 | 1
Hemorrhage pulmonary, nose (Vascular disorders) | 0 | 1
Infection (documented clinically), bladder (urinary) (Infections and infestations) | 0 | 1
Infection (documented clinically), mucosa (Infections and infestations) | 0 | 1
ALT (Metabolism and nutrition disorders) | 0 | 1
AST (Metabolism and nutrition disorders) | 0 | 1
Hyperkalemia (Metabolism and nutrition disorders) | 0 | 2
Hyperglycemia (Metabolism and nutrition disorders) | 0 | 1
Hyperuricemia (Metabolism and nutrition disorders) | 0 | 3
Hypocalcemia (Metabolism and nutrition disorders) | 0 | 1
Hyponatremia (Metabolism and nutrition disorders) | 0 | 1
Cognitive disturbance (Nervous system disorders) | 0 | 1
Pain, muscle (General disorders) | 0 | 1
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 1
Erythema multiforme (Skin and subcutaneous tissue disorders) | 0 | 2

LIMITATIONS AND CAVEATS:
The study was terminated early by the Sponsor due to low accrual. No efficacy analyses were performed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Protocol and PI clinical trial agreements.